CLINICAL TRIAL: NCT00711464
Title: A Dose-response Study of Modafinil Effects on Cognition in Schizophrenia Patients.
Brief Title: Modafinil Effects on Cognition in Schizophrenia Patients
Acronym: InO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Minzenberg, MD, Associate Professor of Clinical Psychiatry, University of California, Davis
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200715868-1
Record Dates: First submitted 2008-07-02; First posted 2008-07-08 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: cognition, pharmacology, memory, attention
MeSH Terms: conditions — Schizophrenia | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 mg (Experimental): modafinil 100 milligrams oral dose
  Interventions: Drug: modafinil (M1, M2, M4)
- 200 mg (Experimental): modafinil 200 mg oral dose
  Interventions: Drug: modafinil (M1, M2, M4)
- 400 mg (Experimental): modafinil 400 mg oral dose
  Interventions: Drug: modafinil (M1, M2, M4)
- Placebo (Placebo Comparator): Single oral placebo capsule
  Interventions: Drug: modafinil (M1, M2, M4)

INTERVENTIONS:
Drug: modafinil (M1, M2, M4) — modafinil 100, 200, and 400 mg oral dose
  Other Names: Provigil

SUMMARY:
Patients with schizophrenia have problems in thinking, known as cognitive dysfunction. This includes many types of cognitive dysfunction, such as in attention, memory and language. These problems may explain why patients with schizophrenia think and act in unusual ways, and often have problems managing aspects of their lives that healthy adults take for granted. Unfortunately, the biochemical aspects of these dysfunctions are presently unknown, and it is not clear whether current psychiatric medications can improve these functions. A recent FDA-approved medication that may improve this function is modafinil. Studies in animals and healthy adults show that this medication can improve many of these cognitive functions. We plan to study the effects of modafinil on these cognitive processes, by giving various doses of this medication to patients before they perform tasks of these cognitive processes. We predict that when patients receive modafinil, they will perform better on a cognitive test, and that these benefits will depend on the dose given.

DETAILED DESCRIPTION:
Schizophrenia is a disorder of cognition. The cognitive deficits of schizophrenia are present at the onset of the disorder, prior to medication exposure, are persistent during periods of remission, and are strongly related to functional outcome. These deficits prominently include prefrontal cortex-dependent functions. While existing medications effectively treat psychotic symptoms, they exhibit modest benefit at best for cognitive dysfunction. Studies of cognition in animal models indicate that the neurotransmitter systems that mediate many cognitive processes are not generally augmented by existing antipsychotic medications. Therefore, advances in the treatment of schizophrenia will require the study of agents with novel pharmacological profiles to establish their potential to remediate cognitive dysfunction.

This study will evaluate the effects of modafinil on the range of cognitive processes known to be disturbed in schizophrenia. Modafinil is an FDA-approved medication with a unique pharmacological profile and an increasing range of off-label indications. Its neurochemical effects in animal models include elevation of extracellular dopamine (DA), noradrenaline (NA) and glutamate in the neocortex. This profile is favorable for the enhancement of cognitive processes. These neurochemical effects also appear to be selective for cortical versus subcortical brain regions, suggesting that modafinil may have minimal effects on psychotic symptoms, or extrapyramidal, autonomic and hormonal side effects. In addition, it differs from amphetamine in structure, neurochemical profile and behavioral effects, with a lower risk of addictive or cerebrovascular effects. Recent studies in animal models, healthy adults and adults with psychiatric and neurological disorders indicate that modafinil improves prefrontal cognitive functions. This suggests that modafinil is a leading candidate for the treatment of cognitive dysfunction in schizophrenia. We aim to test modafinil effects on the remediation of deficits in cognition in individuals with schizophrenia. We will vary the dose within each participant to evaluate dose-response relationships, and directly compare cognition outcome measures for sensitivity to drug effects.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18-54
* diagnosis of schizophrenia or schizoaffective disorder, or healthy with no personal or family history of mental illness
* able to provide informed consent

Exclusion Criteria:

* history of significant head injury or other neurological illness
* active psychiatric illness requiring significant acute care
* significant intellectual impairment (e.g. standardized full-scale IQ < 70)
* history of medical illness or treatment that is associated with significant increase in risk from modafinil treatment (e.g. cardiac disease)
* significant active substance abuse
* active pregnancy
* active treatment with medications that have drug interactions with modafinil

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Minzenberg, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis School of Medicine, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: modafinil 100 milligrams oral dose, 200 milligrams oral dose, 400 milligrams oral dose, and placebo, in randomly sequenced dosing periods.
Period: Overall Study
Arm/Group | All Participants
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: modafinil (M1, M2, M4): modafinil 100, 200, and 400 mg oral dose, and placebo, in random sequence.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Performance
Description: Percent Accuracy on high-control (i.e. difficult) condition on test of cognitive control
Time Frame: 3-5 hours
Measure: Mean (Standard Deviation); unit: percentage correct of all trials
Arm/Group | 100 mg | 200 mg | 400 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29 | 29
percentage correct of all trials | 76.7 (22.8) | 75.5 (26.8) | 67.2 (33.2) | 77.1 (26.3)

2. Secondary Outcome: Systolic Blood Pressure
Description: systolic blood pressure in mm Hg
Time Frame: 3-5 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 100 mg | 200 mg | 400 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29 | 29
mm Hg | 109 (16) | 112 (14) | 116 (16) | 111 (10)

3. Secondary Outcome: Heart Rate
Description: beats per minute
Time Frame: 3-5 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 100 mg | 200 mg | 400 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29 | 29
beats per minute | 74 (10) | 81 (12) | 86 (16) | 76 (12)

ADVERSE EVENTS:
Time Frame: 6 hours post-dose on treatment days
Arm/Group | 100 mg | 200 mg | 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes